CLINICAL TRIAL: NCT07129512
Title: Clipless Ultrasonic Energy-based Hemostasis Versus Conventional Clipping Hemostasis in Laparoscopic Colorectal Surgery: A Pilot Study
Brief Title: Ultrasonic Versus Conventional Clipping Hemostasis in Laparoscopic Colorectal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2023-1029
Record Dates: First submitted 2024-07-03; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Adenocarcinoma of the Colon
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is a prospective, randomized, single-center study comparing clipless ultrasonic energy-based hemostasis versus conventional clipping hemostasis in performing laparoscopic colectomy. The study subjects will be randomly assigned to: 1. clipless ultrasonic energy-based hemostasis 2. conventional clipping hemostasis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clipless ultrasonic energy-based hemostasis (Experimental): In this group, the vessel ligation and dissection is performed using an ultrasonic scalpel with advanced hemostasis mode.
  Interventions: Procedure: Intracorporeal anastomosis
- Conventional clipping hemostasis (Active Comparator): In this group, the vessel ligation and dissection is performed using a monopolar energy device and surgical clips.
  Interventions: Procedure: Extracorporeal anastomosis

INTERVENTIONS:
Procedure: Intracorporeal anastomosis — In this group, the vessel ligation and dissection is performed using an ultrasonic scalpel with advanced hemostasis mode.
  Arms: Clipless ultrasonic energy-based hemostasis
Procedure: Extracorporeal anastomosis — In this group, the vessel ligation and dissection is performed using a monopolar energy device and surgical clips.
  Arms: Conventional clipping hemostasis

SUMMARY:
INTRODUCTION Colorectal cancer rates are rising, with surgery emphasizing radical resection and vessel ligation. Conventional methods using clips pose risks of bleeding and complications. Ultrasonic scalpels offer a safer alternative, approved for various surgeries, but their efficacy in colorectal cancer surgery needs prospective validation.

STUDY OBJECTIVE Study compares safety/efficacy of clipless vs. clip-type hemostasis using ultrasonic scalpel in colorectal surgery, focusing on post-op bleeding frequency, intraoperative bleed, drainage, hospital stay.

STUDY DESIGN This study is a prospective, randomized, single-center study comparing clipless ultrasonic energy-based hemostasis versus conventional clipping hemostasis in performing laparoscopic colectomy. The study's experimental group undergoes surgery with an ultrasonic scalpel, while the control group receives treatment with a monopolar energy device and clips. Allocation to groups, using a 1:1 ratio, is randomized via a computerized table by a blinded coordinator, immediately post-anesthesia. Principal investigators and administrators remain blinded throughout the study.

STUDY POPULATION

1. Screening A detailed review of the medical records will be performed to assess inclusion/exclusion criteria for all subjects who have been diagnosed with colonic adenocarcinoma and are subject to a colectomy procedure.

All patients who are eligible, meet the inclusion and none of the exclusion criteria of this study, will be offered enrollment into the study at each site.

RISK ANALYSIS The surgical procedure, postoperative care, and follow-up will be the same for the experitmental and control groups in this study. The use of the ultrasonic scalpel alone may prevent complications such as clip-induced intestinal obstruction, infection, bleeding from clip dislodgement, bile leakage, and infection, but there is no additional benefit for other subjects. The risk of bleeding when ligating vessels with an ultrasonic scalpel has been demonstrated to be safe in retrospective studies for vessels 7 mm or less (8-17). Vessels larger than 7 mm are ligated using surgical clips because the safety of ligation with the ultrasound scalpel has not been studied. Based on the reported safety of this method of ligation, the risks do not outweigh the benefits when analyzed in the aggregate.

QUALIFICATION OF PARTICIPATING SURGEONS

1. Surgical procedure

   * Laparoscopic surgery: Surgery for colorectal cancer consists of ligating blood vessels to the lesion, detaching or mobilizing the colon, and resecting and anastomosing the bowel.
   * Clipless ultrasound energy-based hemostasis arm: the ultrasound scalpel is used to dissect and ligate the vessel, but clips are used for vessels larger than 7 mm in diameter. If there is significant bleeding during the procedure, surgical clips and hemostatic agents may be used for patient safety at the discretion of the surgeon.
   * Control arm: a combination of monopolar cautery and surgical clips will be used for vascular ligation and lymph node dissection.
2. Procedure standardization and qualification procedure This study is about laparoscopic surgery for colorectal cancer and all surgeries will be performed by surgeons with at least 100 laparoscopic colorectal cancer surgeries.

STATISTICAL ANALYSIS This study compares the frequency of postoperative bleeding between clipless and clip-type ultrasound energy hemostasis in laparoscopic colorectal cancer surgery, assuming that there will be deviations from randomization, such as switching of surgical groups after randomization or additional vessel ligation with clips during or after surgery, we will perform a per-protocol analysis.

The missing values of postoperative bleeding, intraoperative blood loss, intraoperative blood transfusion, and conversion to laparotomy are assumed to be none, and the missing values of postoperative drainage tube hematocrit and drainage tube triglycerides are converted to the mean values of the same group. Outliers will be retained without replacement for intraoperative blood loss, operative time, maximum postoperative plasma hemoglobin decline, and total drainage volume within 5 days postoperatively.

For Type 1 errors, the frequency of postoperative intra-abdominal bleeding in the control group will be analyzed during data safety monitoring every 50 cases to ensure that it is less than 0.5-4.5% according to the literature.

DETAILED DESCRIPTION:
STUDY METHODS

1. Ethical committee approval The study protocol, patient informed consent form and other required study documentation will be reviewed and approved by an institutional review board or any other authority body, prior to study start-up.
2. Study duration and enrollment The total study duration will be approximately 5 years. Study enrollment will take approximately 18 months. The study subjects will have a short-term follow-up at 30 days after surgery. Surveillance will be performed according to standard follow-up guideline after colorectal cancer surgery.
3. Randomization A computerized random number table allocating subjects to treatment and control groups in a 1:1 ratio will be administered by a clinically blinded study coordinator, and allocation will be performed immediately after anesthesia in the operating room on the day of surgery. The principal investigator and administrator will be blinded.
4. Data collection Data will be collected at baseline, post-operative, discharge and 1 month. A screening log will be maintained at each site during the enrollment period, in which all patients eligible for the trial shall be identified. This will be maintained to ensure no patient selection bias occurs within a center or by a surgeon.
5. Informed Consent Using the study-specific, IRB approved, informed consent form, information pertinent to this study will be provided to the subjects in writing and in their native, non-technical, language. The consent form will include a description of the study and its purpose, potential benefits, potential risks, site contact information, and all other elements required of an informed consent.

   Subjects are required to voluntarily sign the informed consent form before any study-specific procedure is performed. The Investigator and/or his/her authorized designee, trained on the protocol and performing a consent, will conduct the informed consent process and will answer questions the subjects may have. If the subject agrees to participate, the informed consent form must be signed and dated by the subject or his/her legally authorized representative prior to enrollment in the study and separately signed and dated by the person taking consent. Only subjects who have signed the study informed consent will be included in the study.
6. Withdrawal and discontinuation The subject's participation in any clinical trial is voluntary. The subject has the right to withdraw at any time without penalty or loss of benefit. Study withdrawal means the subject is no longer participating in the study and no further follow-ups will be performed. All subjects that withdraw after informed consent is signed will be evaluated at the time of withdrawal. Every effort will be made to document the subject outcome at the time of withdrawal. The investigator has the right to discontinue subjects from the study at their discretion to ensure wellbeing of the subject. The reasons for withdrawal shall be documented.

STUDY METHODS

1. Ethical committee approval The study protocol, patient informed consent form and other required study documentation will be reviewed and approved by an institutional review board or any other authority body, prior to study start-up.
2. Study duration and enrollment The total study duration will be approximately 5 years. Study enrollment will take approximately 18 months. The study subjects will have a short-term follow-up at 30 days after surgery. Surveillance will be performed according to standard follow-up guideline after colorectal cancer surgery.
3. Randomization A computerized random number table allocating subjects to treatment and control groups in a 1:1 ratio will be administered by a clinically blinded study coordinator, and allocation will be performed immediately after anesthesia in the operating room on the day of surgery. The principal investigator and administrator will be blinded.
4. Data collection Data will be collected at baseline, post-operative, discharge and 1 month. A screening log will be maintained at each site during the enrollment period, in which all patients eligible for the trial shall be identified. This will be maintained to ensure no patient selection bias occurs within a center or by a surgeon.
5. Informed Consent Using the study-specific, IRB approved, informed consent form, information pertinent to this study will be provided to the subjects in writing and in their native, non-technical, language. The consent form will include a description of the study and its purpose, potential benefits, potential risks, site contact information, and all other elements required of an informed consent.

   Subjects are required to voluntarily sign the informed consent form before any study-specific procedure is performed. The Investigator and/or his/her authorized designee, trained on the protocol and performing a consent, will conduct the informed consent process and will answer questions the subjects may have. If the subject agrees to participate, the informed consent form must be signed and dated by the subject or his/her legally authorized representative prior to enrollment in the study and separately signed and dated by the person taking consent. Only subjects who have signed the study informed consent will be included in the study.
6. Withdrawal and discontinuation The subject's participation in any clinical trial is voluntary. The subject has the right to withdraw at any time without penalty or loss of benefit. Study withdrawal means the subject is no longer participating in the study and no further follow-ups will be performed. All subjects that withdraw after informed consent is signed will be evaluated at the time of withdrawal. Every effort will be made to document the subject outcome at the time of withdrawal. The investigator has the right to discontinue subjects from the study at their discretion to ensure wellbeing of the subject. The reasons for withdrawal shall be documented.

STUDY METHODS

1. Ethical committee approval The study protocol, patient informed consent form and other required study documentation will be reviewed and approved by an institutional review board or any other authority body, prior to study start-up.
2. Study duration and enrollment The total study duration will be approximately 5 years. Study enrollment will take approximately 18 months. The study subjects will have a short-term follow-up at 30 days after surgery. Surveillance will be performed according to standard follow-up guideline after colorectal cancer surgery.
3. Randomization A computerized random number table allocating subjects to treatment and control groups in a 1:1 ratio will be administered by a clinically blinded study coordinator, and allocation will be performed immediately after anesthesia in the operating room on the day of surgery. The principal investigator and administrator will be blinded.
4. Data collection Data will be collected at baseline, post-operative, discharge and 1 month. A screening log will be maintained at each site during the enrollment period, in which all patients eligible for the trial shall be identified. This will be maintained to ensure no patient selection bias occurs within a center or by a surgeon.
5. Informed Consent Using the study-specific, IRB approved, informed consent form, information pertinent to this study will be provided to the subjects in writing and in their native, non-technical, language. The consent form will include a description of the study and its purpose, potential benefits, potential risks, site contact information, and all other elements required of an informed consent.

   Subjects are required to voluntarily sign the informed consent form before any study-specific procedure is performed. The Investigator and/or his/her authorized designee, trained on the protocol and performing a consent, will conduct the informed consent process and will answer questions the subjects may have. If the subject agrees to participate, the informed consent form must be signed and dated by the subject or his/her legally authorized representative prior to enrollment in the study and separately signed and dated by the person taking consent. Only subjects who have signed the study informed consent will be included in the study.
6. Withdrawal and discontinuation The subject's participation in any clinical trial is voluntary. The subject has the right to withdraw at any time without penalty or loss of benefit. Study withdrawal means the subject is no longer participating in the study and no further follow-ups will be performed. All subjects that withdraw after informed consent is signed will be evaluated at the time of withdrawal. Every effort will be made to document the subject outcome at the time of withdrawal. The investigator has the right to discontinue subjects from the study at their discretion to ensure wellbeing of the subject. The reasons for withdrawal shall be documented.

STUDY METHODS

1. Ethical committee approval The study protocol, patient informed consent form and other required study documentation will be reviewed and approved by an institutional review board or any other authority body, prior to study start-up.
2. Study duration and enrollment The total study duration will be approximately 5 years. Study enrollment will take approximately 18 months. The study subjects will have a short-term follow-up at 30 days after surgery. Surveillance will be performed according to standard follow-up guideline after colorectal cancer surgery.
3. Randomization A computerized random number table allocating subjects to treatment and control groups in a 1:1 ratio will be administered by a clinically blinded study coordinator, and allocation will be performed immediately after anesthesia in the operating room on the day of surgery. The principal investigator and administrator will be blinded.
4. Data collection Data will be collected at baseline, post-operative, discharge and 1 month. A screening log will be maintained at each site during the enrollment period, in which all patients eligible for the trial shall be identified. This will be maintained to ensure no patient selection bias occurs within a center or by a surgeon.
5. Informed Consent Using the study-specific, IRB approved, informed consent form, information pertinent to this study will be provided to the subjects in writing and in their native, non-technical, language. The consent form will include a description of the study and its purpose, potential benefits, potential risks, site contact information, and all other elements required of an informed consent.

   Subjects are required to voluntarily sign the informed consent form before any study-specific procedure is performed. The Investigator and/or his/her authorized designee, trained on the protocol and performing a consent, will conduct the informed consent process and will answer questions the subjects may have. If the subject agrees to participate, the informed consent form must be signed and dated by the subject or his/her legally authorized representative prior to enrollment in the study and separately signed and dated by the person taking consent. Only subjects who have signed the study informed consent will be included in the study.
6. Withdrawal and discontinuation The subject's participation in any clinical trial is voluntary. The subject has the right to withdraw at any time without penalty or loss of benefit. Study withdrawal means the subject is no longer participating in the study and no further follow-ups will be performed. All subjects that withdraw after informed consent is signed will be evaluated at the time of withdrawal. Every effort will be made to document the subject outcome at the time of withdrawal. The investigator has the right to discontinue subjects from the study at their discretion to ensure wellbeing of the subject. The reasons for withdrawal shall be documented.

STUDY METHODS

1. Ethical committee approval The study protocol, patient informed consent form and other required study documentation will be reviewed and approved by an institutional review board or any other authority body, prior to study start-up.
2. Study duration and enrollment The total study duration will be approximately 5 years. Study enrollment will take approximately 18 months. The study subjects will have a short-term follow-up at 30 days after surgery. Surveillance will be performed according to standard follow-up guideline after colorectal cancer surgery.
3. Randomization A computerized random number table allocating subjects to treatment and control groups in a 1:1 ratio will be administered by a clinically blinded study coordinator, and allocation will be performed immediately after anesthesia in the operating room on the day of surgery. The principal investigator and administrator will be blinded.
4. Data collection Data will be collected at baseline, post-operative, discharge and 1 month. A screening log will be maintained at each site during the enrollment period, in which all patients eligible for the trial shall be identified. This will be maintained to ensure no patient selection bias occurs within a center or by a surgeon.
5. Informed Consent Using the study-specific, IRB approved, informed consent form, information pertinent to this study will be provided to the subjects in writing and in their native, non-technical, language. The consent form will include a description of the study and its purpose, potential benefits, potential risks, site contact information, and all other elements required of an informed consent.

   Subjects are required to voluntarily sign the informed consent form before any study-specific procedure is performed. The Investigator and/or his/her authorized designee, trained on the protocol and performing a consent, will conduct the informed consent process and will answer questions the subjects may have. If the subject agrees to participate, the informed consent form must be signed and dated by the subject or his/her legally authorized representative prior to enrollment in the study and separately signed and dated by the person taking consent. Only subjects who have signed the study informed consent will be included in the study.
6. Withdrawal and discontinuation The subject's participation in any clinical trial is voluntary. The subject has the right to withdraw at any time without penalty or loss of benefit. Study withdrawal means the subject is no longer participating in the study and no further follow-ups will be performed. All subjects that withdraw after informed consent is signed will be evaluated at the time of withdrawal. Every effort will be made to document the subject outcome at the time of withdrawal. The investigator has the right to discontinue subjects from the study at their discretion to ensure wellbeing of the subject. The reasons for withdrawal shall be documented.

STUDY METHODS

1. Ethical committee approval The study protocol, patient informed consent form and other required study documentation will be reviewed and approved by an institutional review board or any other authority body, prior to study start-up.
2. Study duration and enrollment The total study duration will be approximately 5 years. Study enrollment will take approximately 18 months. The study subjects will have a short-term follow-up at 30 days after surgery. Surveillance will be performed according to standard follow-up guideline after colorectal cancer surgery.
3. Randomization A computerized random number table allocating subjects to treatment and control groups in a 1:1 ratio will be administered by a clinically blinded study coordinator, and allocation will be performed immediately after anesthesia in the operating room on the day of surgery. The principal investigator and administrator will be blinded.
4. Data collection Data will be collected at baseline, post-operative, discharge and 1 month. A screening log will be maintained at each site during the enrollment period, in which all patients eligible for the trial shall be identified. This will be maintained to ensure no patient selection bias occurs within a center or by a surgeon.
5. Informed Consent Using the study-specific, IRB approved, informed consent form, information pertinent to this study will be provided to the subjects in writing and in their native, non-technical, language. The consent form will include a description of the study and its purpose, potential benefits, potential risks, site contact information, and all other elements required of an informed consent.

   Subjects are required to voluntarily sign the informed consent form before any study-specific procedure is performed. The Investigator and/or his/her authorized designee, trained on the protocol and performing a consent, will conduct the informed consent process and will answer questions the subjects may have. If the subject agrees to participate, the informed consent form must be signed and dated by the subject or his/her legally authorized representative prior to enrollment in the study and separately signed and dated by the person taking consent. Only subjects who have signed the study informed consent will be included in the study.
6. Withdrawal and discontinuation The subject's participation in any clinical trial is voluntary. The subject has the right to withdraw at any time without penalty or loss of benefit. Study withdrawal means the subject is no longer participating in the study and no further follow-ups will be performed. All subjects that withdraw after informed consent is signed will be evaluated at the time of withdrawal. Every effort will be made to document the subject outcome at the time of withdrawal. The investigator has the right to discontinue subjects from the study at their discretion to ensure wellbeing of the subject. The reasons for withdrawal shall be documented.

STUDY METHODS

1. Ethical committee approval The study protocol, patient informed consent form and other required study documentation will be reviewed and approved by an institutional review board or any other authority body, prior to study start-up.
2. Study duration and enrollment The total study duration will be approximately 5 years. Study enrollment will take approximately 18 months. The study subjects will have a short-term follow-up at 30 days after surgery. Surveillance will be performed according to standard follow-up guideline after colorectal cancer surgery.
3. Randomization A computerized random number table allocating subjects to treatment and control groups in a 1:1 ratio will be administered by a clinically blinded study coordinator, and allocation will be performed immediately after anesthesia in the operating room on the day of surgery. The principal investigator and administrator will be blinded.
4. Data collection Data will be collected at baseline, post-operative, discharge and 1 month. A screening log will be maintained at each site during the enrollment period, in which all patients eligible for the trial shall be identified. This will be maintained to ensure no patient selection bias occurs within a center or by a surgeon.
5. Informed Consent Using the study-specific, IRB approved, informed consent form, information pertinent to this study will be provided to the subjects in writing and in their native, non-technical, language. The consent form will include a description of the study and its purpose, potential benefits, potential risks, site contact information, and all other elements required of an informed consent.

   Subjects are required to voluntarily sign the informed consent form before any study-specific procedure is performed. The Investigator and/or his/her authorized designee, trained on the protocol and performing a consent, will conduct the informed consent process and will answer questions the subjects may have. If the subject agrees to participate, the informed consent form must be signed and dated by the subject or his/her legally authorized representative prior to enrollment in the study and separately signed and dated by the person taking consent. Only subjects who have signed the study informed consent will be included in the study.
6. Withdrawal and discontinuation The subject's participation in any clinical trial is voluntary. The subject has the right to withdraw at any time without penalty or loss of benefit. Study withdrawal means the subject is no longer participating in the study and no further follow-ups will be performed. All subjects that withdraw after informed consent is signed will be evaluated at the time of withdrawal. Every effort will be made to document the subject outcome at the time of withdrawal. The investigator has the right to discontinue subjects from the study at their discretion to ensure wellbeing of the subject. The reasons for withdrawal shall be documented.

ELIGIBILITY:
Inclusion Criteria:

* Adults 19 to 80 years of age
* Patients with histologically confirmed pathologic adenocarcinoma of the colon
* Patients with an ECOG score between 0 and 2
* Patients with a preoperative ASA score of I to III
* Patients without a history of surgery for abdominal malignancies
* Patients with no history of anticoagulation prior to surgery
* Patients who understand the study process and treatment plan and are able to complete the informed consent form themselves

Exclusion Criteria:

* Patients with an ASA score of 4 or higher
* People with blood clotting disorders such as liver cirrhosis, end-stage renal failure, or hematologic disorders
* Pregnant women
* Mentally ill patients who have difficulty giving informed consent
* Preoperative blood hemoglobin (Hb) less than 7 g/dL
* Patients taking anticoagulants before or after surgery
* Patients who have undergone emergency surgery
* Patients who are unable to be followed up on an outpatient basi
* No Informed consent

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-24 (Estimated)

PRIMARY OUTCOMES:
Frequency of postoperative intra-abdominal bleeding with Clavien-Dindo grade II or higher | within 30 postoperative days
  Evaluation of the presence of intra-abdominal bleeding after surgery for Clavien-Dindo grade II or greater is considered positive if any of the following are satisfied within postoperative 30 days
  1. Blood transfusion was performed because of suspected intra-abdominal bleeding.
  2. A contrast-enhanced abdominal pelvic tomogram performed for suspected intra-abdominal hemorrhage demonstrates contrast leakage or the presence of a hemoperitoneum.
  3. Angiographic thromboembolization for intra-abdominal bleeding.
  4. Reoperation for intra-abdominal bleeding.

SECONDARY OUTCOMES:
Intraoperative blood loss (estimated blood loss, ml) | intraoperative
  Volume of blood lost during the surgical procedure, estimated by the anesthesiologist based on suction canister volume and surgical field assessment, excluding irrigation fluid.
intraoperative blood transfusion | intraoperative
  Whether the participant received any transfusion of packed red blood cells, fresh frozen plasma, or platelets during surgery, as documented in anesthesia and operative records.
conversion to laparotomy | intraoperative
  Whether laparoscopic surgery was converted to open laparotomy for any reason, including uncontrolled bleeding, poor exposure, or intraoperative injury.
operative time | intraoperative
  Total duration of the surgical procedure from skin incision to wound closure, recorded in operative notes.
postoperative plasma hemoglobin maximum decrease (mg/dL) | 5 days
  Largest drop in hemoglobin concentration compared with the preoperative baseline, measured from postoperative blood samples.
total drainage tube volume (ml) within 5 days postoperatively | 5 days
  Cumulative drainage output from the indwelling drain over the first 5 postoperative days, measured daily and summed.
postoperative drainage tube hematocrit (Hct) (maximum value) | 5 days
  Highest hematocrit value measured from drainage fluid samples during the first 5 postoperative days.
drainage tube triglyceride (TG) (maximum value) | 5 days
  Highest triglyceride concentration measured from drainage fluid samples during the first 5 postoperative days.
complications within 30 days postoperatively | 30 days
  Any postoperative adverse event graded using the Clavien-Dindo classification. Report both overall complications (any grade) and clinically significant complications (grade ≥ II). Data obtained from inpatient records and outpatient follow-up within 30 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Colon and Rectal Surgery, Department of Surgery, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No